CLINICAL TRIAL: NCT04004338
Title: Patient Related Outcomes in Real Life Prospective Follow up Study: Carfilzomib in Combination for the Treatment of RR MM
Brief Title: Carfilzomib in Combination for the Treatment of RR MM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Black Sea Hematology Association (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20187462
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Carfilzomib; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Kyprolis — Patients receiving kyprolis (carfilzomib)

SUMMARY:
Carfilzomib is approved in Turkey for the treatment of adult relapsed multiple myeloma patients who have received at least one prior treatment. It is approved for use in combination with lenalidomide and dexamethasone (KRd) in and with dexamethasone alone (Kd). The purpose of this study is to describe contemporary, real-world patterns of patient characteristics, clinical disease presentation, prior therapeutic regimen chosen, and clinical outcomes in participants with relapsed/refractory (R/R) multiple myeloma (MM) who receive Carfilzomib combination treatment. Real-world evidence is crucial to understand how carfilzomib-based regimens are used in practice and in relation to local prescribing information.

This is a prospective, non-interventional, observational study.

The study population will include patients with relapsed/refractory MM who have received 1 to 3 prior lines of therapy with documented data in the medical record regarding diagnosis (month and year), the regimens used in 1st, 2nd, and 3rd line as applicable, whether stem cell transplant was part of 1st, 2nd, and 3rd line of therapy at participating clinical sites in Turkey.

DETAILED DESCRIPTION:
Carfilzomib is approved in Turkey for the treatment of adult relapsed multiple myeloma patients who have received at least one prior treatment. It is approved for use in combination with lenalidomide and dexamethasone (KRd) in and with dexamethasone alone (Kd). The purpose of this study is to describe contemporary, real-world patterns of patient characteristics, clinical disease presentation, prior therapeutic regimen chosen, and clinical outcomes in participants with relapsed/refractory (R/R) multiple myeloma (MM) who receive Carfilzomib combination treatment. Real-world evidence is crucial to understand how carfilzomib-based regimens are used in practice and in relation to local prescribing information.

This is a prospective, non-interventional, observational study.

The study population will include patients with relapsed/refractory MM who have received 1 to 3 prior lines of therapy with documented data in the medical record regarding diagnosis (month and year), the regimens used in 1st, 2nd, and 3rd line as applicable, whether stem cell transplant was part of 1st, 2nd, and 3rd line of therapy at participating clinical sites in Turkey.

For the primary and secondary objectives, analyses will be descriptive and include estimations; no formal hypotheses will be tested.

The study will enroll 300 participants. This multi-center trial will be conducted in Turkish Hematology clinics. The overall time to participate in this study is 12 months. Participants will be evaluated and followed-up for a period of at 12 months, until death, are lost to follow-up, or the end of the study, whichever comes first.

All hematology centers that treat MM will be eligible for participation in this study; it is likely that most participating sites will be academic institutions and/or large specialized hematology centers that treat a relatively high volume of patients with MM. It is estimated that a selection of 20 sites will be required to achieve a target of 300 patients in this study.

It is estimated that 300 RR MM patients receiving treatment will be included in the study. It is expected that this sample size will provide acceptable precision around the estimates of the primary and secondary study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Relapsed/refractory MM patients who have received 1 to 3 prior lines of therapy
* Is willing and able to sign informed consent (ICF) to participate
* Patients receiving carfilzomib equal or less than 2 months (≤2 cycles) according to regulatory approvals

Exclusion Criteria:

* Is reporting to a site in this study for a second opinion (consultation only) or participants whose frequency of consult and follow-up are not adequate for case report form (eCRF) completion.
* Is participating in another study (observational or interventional) that prohibits participation in this study.
* Patients receiving carfilzomib more than 2 months (>2 cycles).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients with relapsed/refractory MM who have received 1 to 3 prior lines of therapy with documented data in the medical record regarding diagnosis (month and year), the regimens used in 1st, 2nd, and 3rd line as applicable, whether stem cell transplant was part of 1st, 2nd, and 3rd line of therapy at participating clinical sites in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-14 (Actual); Primary Completion 2021-04-14 (Estimated); Study Completion 2021-04-14 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months
  Treatment initiation to progression or death

SECONDARY OUTCOMES:
Dyspnea Frequency | 24 months
  Grading according to CTCAE v4.02

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Turgut, Prof, Principal Investigator — 19 Mayıs University Faculty of Medicine
Locations (1):
- 19 Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided